CLINICAL TRIAL: NCT01819753
Title: Assessment of the Effects of Access Count in Percutaneous Nephrolithotomy on Renal Functions by Technetium-99M-Dimercaptosuccinic Acid Scintigraphy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Abdullah Demirtas, Assistant Professor., MD, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DMSAPCNL
Record Dates: First submitted 2013-03-25; First posted 2013-03-28 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2013-03

CONDITIONS: Renal Parenchymal Loss After the Percutaneous Nephrolithotomy
Keywords: percutaneous nephrolithotomy; urinary Stones; 99m-Technetium-Dimercaptosuccinic Acid
MeSH Terms: conditions — Urinary Calculi | interventions — Nephrolithotomy, Percutaneous

ARMS (2):
- Single access (Active Comparator): It was performed only single access standard PCNL in this group.
  Interventions: Procedure: Percutaneous nephrolithotomy
- Multiple access (Active Comparator): It was performed multiple access standard PCNL in this group
  Interventions: Procedure: Percutaneous nephrolithotomy

INTERVENTIONS:
Procedure: Percutaneous nephrolithotomy — The procedure is done under general anesthesia in the supine position. A Retrograde pyelogram is done to locate the stone in the kidney. With a small incision in the flank, the percutaneous nephrolithotomy (PCN) needle is passed into the pelvis of the kidney. The position of the needle is confirmed by fluoroscopy. A guide wire is passed through the needle into the pelvis. The needle is then withdrawn with the guide wire still inside the pelvis. Over the guide wire the dilators are passed and a working sheath is introduced. A nephroscope is then passed inside and stones are taken out.

SUMMARY:
In this study 37 patients who had undergone percutaneous nephrolithotomy were included. Preoperative DMSA scans were performed a day before the surgery, whereas postoperative scans were randomized by evaluating them before (n=25) and after (n=12) the 6th postoperative month. A DMSA scan was read by using a technique that divides both kidneys into three paired poles. In this way functional changes were investigated in the renal units. Twenty six of 37 cases underwent percutaneous nephrolithotomy with a single access site and 11 with multiple access sites. When each of the poles of a kidney was admitted as a surgical unit separately, there were 51 units.

DETAILED DESCRIPTION:
Total 37 patients who had undergone PCNL were included between June 2007-June 2009. All patients were evaluated routinely with physical examination, complete blood count (CBC), blood urine nitrogen (BUN), creatinine levels, and urinalysis. None of the patients had experienced pyelonephritis, and none had a solitary kidney, renal ectopy or history of any other urinary abnormality. At least one of the following techniques; namely computed tomography (CT), intravenous urography or ultrasonography, was preferred routinely before surgery in order to visualize the urinary system. Unilateral PCNL was performed in all patients. Postoperative CBC and BUN creatine levels were repeated.

Preoperative DMSA scans were performed a day before the surgery, whereas postoperative scans were randomized to indicate early and late term. The aim of randomization was to determine an optimal time for assessing patients. A DMSA scan was read by using a technique that divides both kidneys into three paired poles. In addition the uptake of all opposite poles was measured together and calculated as a percentage value separately (Figure-1), e.g., the two upper poles' uptake was measured together as if they were renal units and each poles' own portion in this total uptake was declared separately as a percentage. How the differential functions were changed between the sides undergoing PCNL and the opposite sides, as well the changes before and 6 months after surgery are manifested by using these parameters.

Twenty six of 37 cases underwent PCNL with a single access site (70.3%) and 11 separately with multiple accesses (29.7%). When each of the poles of a kidney was considered as a surgical unit, there were 51 units. In this manner the functional change of a unit would show the surgical trauma inflicted on the poles by PCNL access.

ELIGIBILITY:
Inclusion Criteria:

- Patients with renal stones which was bigger than 2cm.

Exclusion Criteria:

* Patients with acute urinary tract infection,
* Patients with bleeding disorder,
* Patients with chronic renal failure,
* Patients with solitary kidney, renal ectopy or history of any other urinary abnormality.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2007-06; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Renal parenchymal function on DMSA before and after percutaneous nephrolithotomy. | six months
  Preoperative DMSA scans were performed a day before percutaneous nephrolithotomy.How the differential functions with DMSA scans were changed between the sides undergoing PCNL and the opposite sides, as well the changes before and 6 months after surgery are manifested by using these parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Demirtaş, Assistant Prof., MD, Study Chair — Department of Urology, Erciyes University Faculty of Medicine, Kayseri, Turkey.
Locations (1):
- Erciyes University Faculty of Medicine., Kayseri, Turkey (Türkiye)